CLINICAL TRIAL: NCT06461884
Title: Combined Effects of Percussion With Diaphragmatic Breathing Exercises on Airway Clearance in Elderly Pneumonia Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0379
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Pneumonia
Keywords: CAP, Diaphragmatic breathing, Percussion and Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: The group A will receive percussions and diaphragmatic breathing with 1 session a day for 3 days in a week for 4 weeks. In this way total 12 sessions will be given to the patients. And group B will receive only diaphragmatic breathing with 1 session a day for total 3 days in a week for 4 weeks
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Percussions (Experimental): Group A: Percussions and diaphragmatic breathing exercise will be performed with 1 session a day for total 3 days in a week for 4 weeks
  Interventions: Other: Percussions
- Diaphragmatic breathing exercise (Experimental): Group B: Diaphragmatic breathing exercise will be performed with 1 session a day for total 3 days in a week for 4 weeks
  Interventions: Other: , Diaphragmatic breathing exercise

INTERVENTIONS:
Other: Percussions — Group A: Percussions and diaphragmatic breathing exercise will be performed with 1 session a day for total 3 days in a week for 4 weeks
  Arms: Percussions
Other: , Diaphragmatic breathing exercise — Group B: Diaphragmatic breathing exercise will be performed with 1 session a day for total 3 days in a week for 4 weeks
  Arms: Diaphragmatic breathing exercise

SUMMARY:
The group A will receive percussions and diaphragmatic breathing with 1 session a day for 3 days in a week for 4 weeks. In this way total 12 sessions will be given to the patients. And group B will receive only diaphragmatic breathing with 1 session a day for total 3 days in a week for 4 weeks. By this intervention procedure, I will find out the effects of these techniques on airway clearance of the pneumonia patients, their effect on the quality of life and on Dyspnea. For this I will use 4 tool questionnaires that are 1-BCSS, 2- Modified Borg Dyspnea scale, 3-Rate of perceived exertion scale, 4- Health-related Quality of Life-14. BCSS will be used to assess breathlessness, cough and sputum retention. Modified Borg Dyspnea scale is 0-10 rated numerical scale used to measure Dyspnea. RPE is a way to measure the level of exertion a person feels during physical activity. HRQOL-14 will assess the quality of life of the pneumonia patients.

DETAILED DESCRIPTION:
It will be a randomized clinical trial. And the data will be conducted from Mayo Hospital Lahore. Convenient sampling technique will be applied on patients according to the inclusion criteria. Patients will be allocated through simple random sampling into group A and group B to collect data. For this purpose, I will divide my sample size into two groups. The group A will receive percussions and diaphragmatic breathing with 1 session a day for 3 days in a week for 4 weeks. In this way total 12 sessions will be given to the patients. And group B will receive only diaphragmatic breathing with 1 session a day for total 3 days in a week for 4 weeks. By this intervention procedure, I will find out the effects of these techniques on airway clearance of the pneumonia patients, their effect on the quality of life and on Dyspnea. For this I will use 4 tool questionnaires that are 1-BCSS, 2- Modified Borg Dyspnea scale, 3-Rate of perceived exertion scale, 4- Health-related Quality of Life-14. BCSS will be used to assess breathlessness, cough and sputum retention. Modified Borg Dyspnea scale is 0-10 rated numerical scale used to measure Dyspnea. RPE is a way to measure the level of exertion a person feels during physical activity. HRQOL-14 will assess the quality of life of the pneumonia patients. Before and after each session, the primary and secondary outcomes will be measured for both groups. After collecting the data, the data will be analyzed by using SPSS version 25.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 40-60,

  * Both males and females
  * Those patients who will be vitally stable (oxygen saturation, respiratory rate)
  * Pneumonia diagnosed patients (Community Acquired Pneumonia)

Exclusion Criteria:

* Patients with heart disease

  * Patients with neurological disorders such as: Alzheimer, epilepsy, Parkinson disease
  * Patients with orthopedic conditions
  * Other pulmonary complications (atelectasis, diaphragmatic injury, ARDS)

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03-10 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
BCSS | 4 weeks
  BCSS: BCSS is a patient-reported three-item questionnaire for cough, breathlessness and sputum rating on a 5-point Likert scale from 0 (no symptoms) to 4 (severe symptoms).
HRQOL for quality of life | 4 weeks
  One of the many factors frequently investigated in the realm of medical research and treatment is HRQOL. It covers a broad spectrum of man experience, contains how we operate and how we perceive illness. The World Health Organization defines health as a condition of whole physical, intellectual, and interpersonal well-being and not just the absence of disease, which is the foundation for modern interpretations of HRQOL.
Rated Perceived Exertion (RPE) Scale | 4 weeks
  Rate of perceived exertion (RPE) is used to measure how hard your body works during physical activity. It runs from 0 - 10, using numbers to rate how much effort an activity takes. The RPE scale can help you manage exercise intensity and improve cardio training and endurance

CONTACTS AND LOCATIONS:
Overall Officials: Sidra Faisal, PP-DPT, Principal Investigator — Riphah International University
Locations (1):
- Mayo Hospital Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jackson ML, Neuzil KM, Thompson WW, Shay DK, Yu O, Hanson CA, Jackson LA. The burden of community-acquired pneumonia in seniors: results of a population-based study. Clin Infect Dis. 2004 Dec 1;39(11):1642-50. doi: 10.1086/425615. Epub 2004 Nov 8. PMID 15578365
- [Background] Brar NK, Niederman MS. Management of community-acquired pneumonia: a review and update. Ther Adv Respir Dis. 2011 Feb;5(1):61-78. doi: 10.1177/1753465810381518. Epub 2010 Oct 8. PMID 20935033
- [Background] Marchello CS, Ebell MH, Dale AP, Harvill ET, Shen Y, Whalen CC. Signs and Symptoms That Rule out Community-Acquired Pneumonia in Outpatient Adults: A Systematic Review and Meta-Analysis. J Am Board Fam Med. 2019 Mar-Apr;32(2):234-247. doi: 10.3122/jabfm.2019.02.180219. PMID 30850460
- [Background] Miyashita N, Yamauchi Y. Bacterial Pneumonia in Elderly Japanese Populations. Jpn Clin Med. 2018 Jan 3;9:1179670717751433. doi: 10.1177/1179670717751433. eCollection 2018. PMID 29434484